CLINICAL TRIAL: NCT07187934
Title: PROSPECTIVE EVALUATION OF THE IDASCORE ALGORITHM FOR EMBRYO RANKING
Brief Title: EVALUATION OF A FULLY AUTOMATED AI TOOL FOR EMBRYO RANKING
Acronym: PRIDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: PRIDE_2025
Record Dates: First submitted 2025-09-04; First posted 2025-09-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy
Keywords: iDA; AI; embryo ranking; transfer-to-pregnancy; time-lapse

STUDY DESIGN:
Intervention Model Description: Randomisation (1:1) based on a computer-generated randomisation list with block size 10.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Embryologist ranking (No Intervention): Embryologist ranks the embryos according to their appearance
- iDA ranking (Experimental): AI tool ranks embryos based on fully automated analysis of time-lapse images
  Interventions: Device: AI algorithm

INTERVENTIONS:
Device: AI algorithm — iDAScore® is a deep learning-based tool that provides fully automated analysis of embryo time-lapse images. It automatically generates a score (1-9.9) for each embryo in the patient's embryo cohort, which correlates to the likelihood of achieving a fetal heartbeat (clinical pregnancy).
  Other Names: iDAScore
  Arms: iDA ranking

SUMMARY:
This study aims to investigate whether embryo ranking by a fully automated AI tool (iDAScore) results in a similar transfer-to-pregnancy compared to manual embryo ranking by an embryologist. IVF patients who are planned for a freeze-all approach (where all usable embryos are frozen and transferred in later transfer cycles) will be allocated to either the control (ranking by embryologist) or intervention arm (ranking by iDAScore). The frozen embryos will be warmed and transferred one by one, according to their assigned rank. We want to see if the average number of embryo transfers that is needed to achieve a clinical pregnancy (transfer-to-pregnancy) is similar in both groups.

DETAILED DESCRIPTION:
The study population consists of IVF/ICSI patients scheduled for a freeze-all policy on day 5. Inclusion takes place on the day prior to oocyte retrieval, based on predefined inclusion criteria. Embryo culture is performed in an EmbryoScope+ time-lapse incubator. On day 5 of embryo development, the embryologist evaluates the embryos using the Gardner criteria, assessing expansion stage, inner cell mass (ICM), and trophectoderm (TE). All embryos meeting our in-house cryopreservation criteria are vitrified. Embryos not yet meeting the criteria remain in culture and are re-evaluated on day 6. Once at least two blastocysts meet the cryopreservation criteria on day 5 and/or day 6, the patient is randomized in the control or study arm.

In the control group, the embryologist manually ranks all freezable embryos according to the assigned Gardner scores, applying a standard prioritization scheme: day of cryopreservation > expansion stage > TE score > ICM score.

If multiple embryos share the same Gardner score, the embryologist looks at the full morphokinetics to establish a final ranking. The order of warming for subsequent frozen embryo transfer (FET) cycles follows this ranking: the embryo ranked 1 is transferred first. If no clinical pregnancy results, the embryo ranked 2 is transferred in the next FET cycle, and so on.

In the study group, the iDA score is retrieved for each freezable embryo. Embryos are ranked solely based on their iDA score, with the highest score assigned rank 1, and so on. The order of warming for subsequent FET cycles is determined exclusively by this ranking. As in the embryologist group, the embryo ranked 1 is transferred first, followed by rank 2 in case of no clinical pregnancy, and so on.

+/- 10 days after embryo transfer, an hCG blood test is performed. In case of a positive result, the pregnancy is monitored until the 7-week ultrasound, at which the presence of fetal heartbeat confirms a clinical pregnancy. Patients are followed for clinical pregnancy outcomes of FETs performed up to one year after oocyte retrieval, or until the pregnancy outcome of the last available embryo is known.

In both the study and control arm, all procedures follow the standard of care. The only difference between the groups is the method of embryo ranking-and therefore the order in which embryos will be transferred.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing an ICSI/IVF treatment (with donor or own oocytes) that are planned for a 'freeze-all' strategy on day 5
* all types of sperm samples (ejaculated or testicular, fresh or frozen, partner or donor origin)
* Minimum 8 follicles (≥ 12 mm) on last follicular measurement before oocyte retrieval
* 18 ≤ Age ≤ 42 years
* 18 ≤ BMI ≤ 35 kg/m²
* Maximum third IVF/ICSI cycle
* Participants can be included only once in the trial

Exclusion Criteria:

* Embassy patients
* Use of frozen oocytes
* In vitro maturation (IVM) cycles
* Pre-implantation genetic Testing (PGT) cycles
* Proven untreated intra-uterine pathologies (e.g. Asherman syndrome, adenomysosis)
* Endometriosis stage 3/4

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only female participants can undergo an oocyte retrieval.
Enrollment: 1325 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2028-12-11 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Transfer to pregnancy | The patient is followed up for clinical pregnancy outcomes (7-week echo) up until 1 year after the oocyte retrieval date, or until the result of the last available embryo is known.
  Number of embryo transfers performed until a clinical pregnancy is obtained

SECONDARY OUTCOMES:
iDA-embryologist consensus | Embryo ranking is done on day 5 and/or 6 of embryo development and can be immediately compared during ranking.
  In how many cases do iDA and the embryologist prioritize the same embryo for the first embryo transfer?
Embryo prioritization time | Measures the time elapsing between the start and end of embryo prioritisation (range of minutes). Is recorded on day 5 and day 6 of embryo development right after embryo evaluation.
  How long does it take to establish a ranking of all embryos from that cohort?
Cumulative clinical pregnancy rate | Up until 1 year after oocyte retrieval
  Number of oocyte retrievals resulting in at least one clinical pregnancy within 1 year of the oocyte retrieval divided by total number of oocyte retrievals
Clinical pregnancy rate after the first embryo transfer | Clinical pregnancy is determined at the 7 week echo by detection of a fetal heart beat.
  Number of clinical pregnancies divided by number of embryo transfers performed

CONTACTS AND LOCATIONS:
Overall Officials: Julie Praet, M.D., Principal Investigator — Brussels IVF, UZ Brussel
Locations (1):
- Brussels IVF, UZ Brussel, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: iDAScore webpage — https://www.vitrolife.com/our-products/idascore-intelligent-data-analysis-for-embryo-evaluation/